CLINICAL TRIAL: NCT04993781
Title: Electronic Strategies for Tailored Exercise to Prevent FallS
Acronym: eSTEPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nancy Latham, PI, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022P001055
Record Dates: First submitted 2021-06-22; First posted 2021-08-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Falls; Fall Injury; Exercise Self-Efficacy; Falls Self-Efficacy

STUDY DESIGN:
Intervention Model Description: The design is a cluster randomized, parallel group superiority trial with practices stratified by healthcare system and patients nested within practices. The unit of randomization is the practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eSTEPS Clinical Decision Support (Experimental): Use of clinical decision support to assist in exercise-related fall prevention care planning will be compared to usual care.
  Interventions: Behavioral: eSTEPS CDS
- Usual Care (No Intervention): Usual primary care practices regarding exercise-related fall prevention planning

INTERVENTIONS:
Behavioral: eSTEPS CDS — Primary care clinics at Brigham and Women's Hospital will be randomized to receive the eSTEPS CDS or usual care. The University of Texas Medical Branch (UTMB) will be the replication site, with all participating primary care practices receiving the eSTEPS CDS.
  Arms: eSTEPS Clinical Decision Support

SUMMARY:
The objectives of this proposal are to evaluate the eSTEPS CDS (eSTEPS) in a cluster randomized controlled trial. The intervention includes the following: 1) A machine learning-based fall injury risk screening algorithm to improve traditional fall risk screening. 2) Provider BPA and/or Care Gap and Smart Set to provide CDS that helps primary care providers develop a tailored fall prevention exercise plan in the context of a Medicare Wellness Visit and 3) eSTEPS Patient App and exercise tools to provide older patients continued access to their interactive, tailored exercise plan.

DETAILED DESCRIPTION:
This project will use traditional fall risk screening and machine learning approaches to accurately identify older adults at risk for falls. Investigators will then develop CDS that will be implemented into the electronic health record that helps primary care providers and older patients develop a tailored fall prevention exercise plan (eSTEPS). The eSTEPS CDS will be integrated into the widely implemented Epic EHR which will be accessible through the Care Gap and SmartSet to provide actionable CDS within primary care clinic workflows and facilitate the use of CDS with older patients during their annual wellness visit, ensuring that evidence-based recommendations are tailored to patients' preferences. The tailored exercise prescription will also be available through printouts, a website, and an app for use by patients at home. The eSTEPS intervention includes the provider CDS and the patient resources (printouts, website, exercise app) that will support primary care providers and patients with personalized exercise care planning during an annual Medicare Wellness visit. Investigators will conduct a cluster randomized controlled trial in urban primary care clinics to test the efficacy of the eSTEPS CDS intervention. Development of the eSTEPS CDS within the widely adopted Epic Electronic Health Record will support dissemination of evidence for older adults.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Age 65 or above
* Patients enrolled in participating primary care intervention and control practices at MGB or enrolled in participating primary care replication trial intervention practices at UTMB
* Positive screen for fall risk at annual wellness visit

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

- Not community-dwelling (i.e. residents of long-term care facilities, prisoners etc.)

Enrollment in the Subsample for Patient Reported Outcomes (PROs):

A subsample of patients will be recruited and consented to participate in follow-up phone calls and surveys. Additional exclusion criteria for the subsample participants are:

* Unwilling or unable to provide verbal consent
* Not able to participate due to cognitive impairment (i.e., 4 or more errors on the Callahan Cognitive Screen assessment)
* Has a terminal illness or other condition that indicates that the participant is not expected to survive for 1 year, such as receiving hospice or palliative care services.
* Not fluent in spoken English
* Does not have access to a working telephone

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 11945 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
To determine the effect of the eSTEPS intervention on the rate of falls | Up to 23 months
  Falls rate per 100 patient years

SECONDARY OUTCOMES:
To determine the effect of the eSTEPS intervention on falls self-efficacy (fear of falling) | Change from initial assessment to 6 months
  Falls self-efficacy (fear of falling) will be measured using the Modified Falls Efficacy Scale (mFES). This scale assesses confidence with completing a list of activities without falling and contains 14 items each measured on a scale of 0 to 10. 0 means "not confident at all", 5 means "fairly confident", and 10 means "completely confident." he total score is the average of all of the item scores and ranges from zero to ten. A higher score reflects more confidence and less fear of falling. Participants are classified as either fearful (MFES score < 8) or not fearful (MFES greater than or equal to 8). The total score range is 0 to 10.
To determine the effect of the eSTEPS intervention on self-efficacy for exercise | Change from initial visit to 6 months
  Self-efficacy for exercise will be measured using the Self-Efficacy for Exercise (SEE) Scale. This scale consists of nine situations that may affect participation in exercise and ask participants to describe their current level of confidence that they could exercise 3 times a week for 20 minutes each time. 0 means "not confident", 5 means "fairly confident", and 10 means "very confident." The total score for the SEE scale is calculated by taking the numerical ratings for each statement and dividing by number of responses. The score indicates the strength of self-efficacy for exercise expectations. The higher the average score, the greater the participant's self-efficacy for exercise. The total score range is 0 to 10.

OTHER OUTCOMES:
To explore the effect of the eSTEPS intervention on the rate of death | Up to 23 months
  Death
To determine the effect of the eSTEPS intervention the rate of fall injuries | Up to 23 months
  Fractures

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT04993781/ICF_000.pdf